CLINICAL TRIAL: NCT01889524
Title: RADIOAEROSSOL PULMONARY DEPOSiTION USING MESH AND JET NEBULIZERS DURING NONINVASIVE VENTILATION IN NORMAL SUBJECTS: A RANDOMIZED CROSSOVER CLINICAL TRIAL
Brief Title: Radioaerossol Pulmonary Deposition Using Mesh in Normal Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Collaborators: Georgia State University (Other); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Daniella Cunha Brandao, PhD, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: valdecir tese normais
Record Dates: First submitted 2013-06-25; First posted 2013-06-28 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Normal Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NIV plus jet (Active Comparator): Noninvasive ventilation-NIV plus jet nebulizer
  Interventions: Other: Jet nebulizer; Other: Noninvasive ventilation-NIV
- NIV plus Mesh (Experimental): Noninvasive ventilation- NIV plus Mesh nebulizer
  Interventions: Other: Mesh nebulizer; Other: Noninvasive ventilation-NIV

INTERVENTIONS:
Other: Mesh nebulizer — VMN (NIVO, Respironics®, Murrysville, Pennsylvania, USA) with an MMAD of 3.0 µm was placed in the elbow adapter at the mask. Inhalation was performed using diethilene triamine penta-acetic technetium (99mTc-DTPA) with radioactivity of 25 millicuries (Nobre et al., 2007). Both nebulizers were charged with 2.5 mg of salbutamol and 0.25 mg of ipratropium bromide and normal saline solution to complete a fill volume of 3 mL.
  Arms: NIV plus Mesh
Other: Jet nebulizer — The JN (Misty Max, Air Life, Yorba Linda, USA) with a particle MMAD of 5 µm (according to the manufacturer information) was positioned in the circuit using a "T" piece placed between the circuit leak and the mask, and operated with oxygen flow at 8 L/min. Inhalation was performed using diethilene triamine penta-acetic technetium (99mTc-DTPA) with radioactivity of 25 millicuries (Nobre et al., 2007). Both nebulizers were charged with 2.5 mg of salbutamol and 0.25 mg of ipratropium bromide and normal saline solution to complete a fill volume of 3 mL.
  Arms: NIV plus jet
Other: Noninvasive ventilation-NIV — Bilevel positive airway pressure (BiPAP Synchrony, Respironics®, Murrysville, Pennsylvania, USA) was applied through face mask (Comfort Full 2, Respironics®, Murrysville, Pennsylvania, USA) attached with straps and pressure adjusted to12 cmH2O peak inspiratory pressure and 5 cmH2O of expiratory pressure at the beginning of the procedure. Patients were adapted to use NIV before starting measurements, pressures were titrated before reaching the established levels and just after this period masks were fitted using the straps. They were oriented to use a breathing pattern inspiring deeply and exhaling slowing to avoid ventilator-patient asynchrony.

SUMMARY:
In vivo deposition studies of aerosol administration during noninvasive ventilation are scarce in the current literature.

We assessed 10 normal subjects in a crossover study evaluated by pulmonary scintigraphy aiming to compare radiaoaerosol pulmonary index and radioaerosol mass balance in the different compartments (pulmonary and extrapulmonary) of radiotagged aerosol administered using vibrating mesh nebulizers (VMN) and conventional jet nebulizer (JN) during noninvasive ventilation (NIV).

ELIGIBILITY:
Inclusion Criteria:

* No history of lung disease;
* Forced vital capacity (FVC) or forced expiratory volume in the first second (FEV1) higher or equal to 80% from predicted values (Pereira et al., 1992),
* No history of smoking;
* Without respiratory or cardiovascular disease;
* Ability to understand verbal commands;
* Willing to provide signed consent to participate in this study.

Exclusion Criteria:

* Pregnant;
* Were unable to tolerate NIV (Metha and Hill, 2001).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-01; Primary Completion 2012-01 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Radioaerosol deposition index | 4 m
  Inhalation was performed using diethilene triamine penta-acetic technetium (99mTc-DTPA) with radioactivity of 25 millicuries (Nobre et al., 2007). Both nebulizers were charged with 2.5 mg of salbutamol and 0.25 mg of ipratropium bromide and normal saline solution to complete a fill volume of 3 mL. The JN (Misty Max, Air Life, Yorba Linda, USA) with a particle MMAD of 5 µm (according to the manufacturer information) was positioned in the circuit using a "T" piece placed between the circuit leak and the mask, and operated with oxygen flow at 8 L/min. VMN (NIVO, Respironics®, Murrysville, Pennsylvania, USA) with an MMAD of 3.0 µm was placed in the elbow adapter at the mask.

SECONDARY OUTCOMES:
Radioaerosol mass balance in pulmonary and extrapulmonary compartments | 4 m
  the same procedure was performed to analysis deposition in the nebulizer, circuits, inspiratory filter, expiratory filter and face mask. Counts representing stomach were obtained from posterior thorax and corrections for decay of technetium were used during extrapulmonary measurements. The analysis of deposition in pulmonary and extrapulmonary compartments was expressed as a percentage from the cumulative count in each compartment representing the total radioaerosol mass.

CONTACTS AND LOCATIONS:
Overall Officials: Valdecir C Galindo Filho, PhD, Principal Investigator — UFPE
Locations (1):
- Hospital das Clínicas, Recife, Pernambuco, Brazil

REFERENCES:
- [Result] Newman SP, Pitcairn GR, Hirst PH, Rankin L. Radionuclide imaging technologies and their use in evaluating asthma drug deposition in the lungs. Adv Drug Deliv Rev. 2003 Jul 18;55(7):851-67. doi: 10.1016/s0169-409x(03)00081-4. PMID 12842604
- [Result] Nobre ME, Lopes F, Cordeiro L, Marinho PE, Silva TN, Amorim C, Cahalin LP, Dornelas de Andrade A. Inspiratory muscle endurance testing: pulmonary ventilation and electromyographic analysis. Respir Physiol Neurobiol. 2007 Jan 15;155(1):41-8. doi: 10.1016/j.resp.2006.04.005. Epub 2006 May 19. PMID 16713403
- [Derived] Galindo-Filho VC, Ramos ME, Rattes CS, Barbosa AK, Brandao DC, Brandao SC, Fink JB, de Andrade AD. Radioaerosol Pulmonary Deposition Using Mesh and Jet Nebulizers During Noninvasive Ventilation in Healthy Subjects. Respir Care. 2015 Sep;60(9):1238-46. doi: 10.4187/respcare.03667. Epub 2015 Jun 23. PMID 26106207